CLINICAL TRIAL: NCT00079846
Title: Safety and Efficacy Study of Implitapide Compared With Placebo in Patients With Homozygous Familial Hypercholesterolemia (HoFH) on Maximal Concurrent Lipid-Lowering Therapy
Brief Title: Implitapide in Patients With Homozygous Familial Hypercholesterolemia (HoFH) on Maximal Concurrent Lipid-Lowering Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Research Laboratories International (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MRL 2002-001
Record Dates: First submitted 2004-03-17; First posted 2004-03-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-04

CONDITIONS: Familial Hypercholesterolemia
Keywords: Homozygous Familial Hypercholesterolemia (HoFH)
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Homozygous Familial Hypercholesterolemia | interventions — implitapide

INTERVENTIONS:
Drug: Implitapide

SUMMARY:
The purpose of this study is to determine if implitapide, used in conjunction with other lipid-lowering therapies, is safe and effective when compared to placebo in lowering low-density lipoprotein cholesterol (LDL-C) in patients with homozygous familial hypercholesterolemia (HoFH).

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, patients must meet all of the following inclusion criteria:

* be between 8 and 70 years old with a diagnosis of HoFH;
* be stable on and maintain concomitant therapy with hypolipidemic drugs or treatments;
* have an appropriate calculated, fasting LDL-C levels and an appropriate triglyceride (TG) level;
* be male or nonpregnant, nonlactating female;
* give informed consent; and
* meet body weight and height requirements.

Exclusion Criteria:

In order to participate in this study, patients must not meet any of the following exclusion criteria:

* recent myocardial infarction, percutaneous transluminal coronary intervention, coronary artery bypass graft surgery, or cerebrovascular accident;
* uncontrolled hypothyroidism or other uncontrolled endocrine disease;
* known, clinically significant eye abnormalities (e.g., cataracts);
* appropriate serum creatinine phosphokinase levels;
* history of liver disease or liver enzyme levels above appropriate levels;
* alkaline phosphatase above appropriate levels;
* liver cirrhosis and severe liver steatosis;
* clinically significant infection, malignancy, or psychosis;
* use of oral anticoagulants or digoxin, unless the dose has been stable for 4 weeks;
* participation in any other investigational study, including device or observational studies, within 30 days;
* lactating or have a positive serum pregnancy test;
* history of or current drug or alcohol abuse; or
* unwillingness to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the investigator.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (6):
- Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio, United States
- Canada (2):
  - Lipid Clinic and Community Genomic Center, Complexe Hospitalier de la Sagamie, Chicoutimi, Quebec
  - Lipid Research Center, CHUL du CHUQ, Sainte-Foy, Quebec
- Hadassah University Hospital, Jerusalem, Israel
- Academic Medical Center Amsterdam, Amsterdam, Netherlands
- Lipidklinikken - Rikshospitalet, Oslo, Norway